CLINICAL TRIAL: NCT02411058
Title: Attention to Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 819369
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-07

CONDITIONS: Informed and Uninformed Incentives
Keywords: information; incentives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uninformed (Experimental): Condition 1
  Interventions: Behavioral: Uninformed
- Informed about Incentives and Purpose (Experimental): Condition 2
  Interventions: Behavioral: Informed

INTERVENTIONS:
Behavioral: Uninformed — Users will receive 20x their usual incentives for two weeks, but will either receive no emails informing them about the incentive program.
  Arms: Uninformed
Behavioral: Informed — Users will receive 20x their usual incentives for two weeks, and they will receive emails informing them about the incentives (one announcement before the incentives begin, and one email every two days reminding them about the overall incentive program). These emails will contain information about the incentives and the purpose of the incentives. The reminder emails sent every two days, however, will include more information about the overall program incentives to maximize the number of participants who learn about the incentive program at some point.
  Arms: Informed about Incentives and Purpose

SUMMARY:
In this experiment, the investigators will test the effectiveness of a two week 20x incentive multiplier on the investigators' corporate partner's users who are (a) not notified about the incentives in advance, and (b) notified about the incentives and their purpose. The investigators will test which group shows the largest boost in walking during the two week intervention and the most lasting behavior change.

DETAILED DESCRIPTION:
Summary:

In this experiment, the investigators will test the effectiveness of a two week 20x incentive multiplier on AchieveMint users who are (a) not notified about the incentives in advance, and (b) notified about the incentives and their purpose. The investigators will test which group shows the largest boost in walking during the two week intervention and the most lasting behavior change.

Information:

The experimental conditions will vary the type and amount of information about incentives as follows:

* Condition 1 - Uninformed: Users will receive 20x their usual incentives for two weeks, but will receive no emails informing them about the incentive program. (They may find out about incentives through the Achievemint platform.)
* Condition 2 - Informed about Incentives and Purpose: Users will receive 20x their usual incentives for two weeks, and they will receive emails informing them about the incentives (one announcement before the incentives begin, and one email every two days reminding them about the overall incentive program). These emails will contain information about the incentives and the purpose of the incentives. Condition 2 will most closely resemble the "constant" condition in the previous experiment. Roughly the same initial announcement email will go out. The reminder emails sent every two days, however, will include more information about the overall program incentives to maximize the number of participants who learn about the incentive program at some point.

Mock-ups of the email announcements and reminders are shown below.

Incentives:

The investigators' incentives will consist of multipliers for points offered via Achievemint. Since the investigators found in the investigators' last experiment that the constant incentives were the most successful, the investigators will offer these incentives to all treated participants: 20x multipliers for 14 days.

Other details:

The other details of the experiment will be the same as the previous experiment:

* Length of incentives: the investigators will offer incentives for 14 days.
* Post-intervention observation: the investigators will observe all treatment groups for at least 30 days after the intervention.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* top 30 percentiles of active walkers
* To the extent possible, given the investigators' target sample size, the investigators will exclude users who were enrolled in the investigators' previous experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2055 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of steps taken | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Milkman, Ph.D., Principal Investigator — University of Pennsylvania; Bradford Tuckfield, Principal Investigator — University of Pennsylvania; Francesco Gino, Ph.D., Principal Investigator — HBS; Leslie K. John, Ph.D., Principal Investigator — HBS
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States